CLINICAL TRIAL: NCT06540547
Title: Supporting Expectant Mothers With ADHD Through the Transition to Parenthood
Brief Title: Moms Managing Attention-Deficit/Hyperactivity Disorder (ADHD) Study
Acronym: MomMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: YourMomCares Foundation (Unknown)
Responsible Party: Principal Investigator, Heather Joseph, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY23100082
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: ADHD; Parenting
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MomMA Intervention (Experimental)
  Interventions: Behavioral: MomMA Intervention

INTERVENTIONS:
Behavioral: MomMA Intervention — Parents will receive sessions of CBT-based behavioral intervention with components targeted specifically towards expectant parents with ADHD. Treatment will be delivered by therapists embedded in OB care settings. The number and specific content of sessions will be determined based on community partner feedback.

SUMMARY:
The study will develop and test a behavioral program for pregnant individuals with Attention-Deficit/Hyperactivity Disorder (ADHD). This behavioral program will include skills for managing ADHD and related symptoms during pregnancy and after delivery and will be taught by a behavioral therapist in OB care settings.

DETAILED DESCRIPTION:
Treating pregnant individuals with ADHD may improve parent and child wellbeing, parent-child interactions, and psychosocial familial factors to enhance family resilience and reduce prevalence/severity of child mental health disorders. Using the information provided from stakeholder interviews and adaptations of an existing CBT intervention for parents of children with ADHD, the current study will develop the MomMA (Moms Managing ADHD) intervention and implement it via an open clinical trial (n=10 pregnant individuals), delivered by masters-level women's health behavioral therapists. Investigators will examine treatment acceptability, feasibility, and appropriateness, as well as implementation factors (fidelity, adherence, facilitators/barriers) and qualitative data (e.g., feedback interviews). In addition, quantitative data (self-reported symptoms, parenting, and home environment measures; observed parent and child behavior; parent reported child temperament/behavior) will be used to assess parent and child outcomes following the intervention. This mixed-methods model will offer a comprehensive examination of the MomMA intervention and inform a refined intervention model.

ELIGIBILITY:
Inclusion Criteria:

* (1) meet full DSM-5 criteria for ADHD
* (2) are between 20- and 32-weeks of gestation
* (3) speak English
* (4) will deliver at the University of Pittsburgh Medical Center (UPMC) Magee Women's Hospital (MWH)

Exclusion Criteria:

* (1) active substance use disorder
* (2) intellectual disability
* (3) other severe mental illness, including bipolar disorder, psychosis, and major depressive disorder with suicidal ideation or requiring higher level of care (inpatient or partial/intensive outpatient)
* (4) high risk pregnancies requiring transfer of care to Maternal-Fetal Medicine (e.g., maternal cancer, multiples, placenta accreta) and/or fetus known to have a severe congenital condition.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-19 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Acceptability | Post Intervention at 4-month postpartum
  Therapist and participant report of intervention acceptability will be assessed using the 4-item Acceptability of Intervention Measure (AIM), rated from rated from 1 (completely disagree) to 5 (completely agree), with scores greater than or equal to 16 indicating good acceptability.
Intervention Appropriateness | Post Intervention at 4-month postpartum
  Therapist and participant report of intervention appropriateness will be assessed using the 4-item Intervention Appropriateness Measure (IAM), rated from 1 (completely disagree) to 5 (completely agree), with scores greater than or equal to 16 indicating good appropriateness.
Intervention Feasibility | Post Intervention at 4-month postpartum
  Therapist and participant report of intervention feasibility will be assessed using the 4-item Feasibility of Intervention Measure (FIM), rated from 1 (completely disagree) to 5 (completely agree), with scores greater than or equal to 16 indicating good feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Joseph, DO, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Magee Women's Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joseph HM, Khetarpal SK, Wilson MA, Molina BSG. Parent ADHD Is Associated With Greater Parenting Distress in the First Year Postpartum. J Atten Disord. 2022 Jul;26(9):1257-1268. doi: 10.1177/10870547211066488. Epub 2021 Dec 23. PMID 34937412
- [Background] Hamilton D. Epilepsy and army physicians. J R Army Med Corps. 1986 Oct;132(3):178-9. No abstract available. PMID 3783529